CLINICAL TRIAL: NCT02475083
Title: Therapeutic Effect of Virtual Reality in Patients After Stroke
Brief Title: Use of Virtual Reality Games for the Treatment of Balance and Reducing the Occurrence of Falls in Patients After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedreira, Érika, M.D. (Individual)
Responsible Party: Principal Investigator, Érika Pedreira, M.D., Pedreira, Érika, M.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EP-13-RV
Record Dates: First submitted 2015-06-12; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2014-08

CONDITIONS: Stroke
Keywords: Stroke; Virtual reality; Balance; Falls
MeSH Terms: conditions — Stroke | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Reality Group (Experimental): Rehabilitation with virtual reality using games with balance training goal.
  Interventions: Other: Virtual Reality; Other: Conventional
- Conventional Group (Active Comparator): Conventional physiotherapy with exercises for balance training.
  Interventions: Other: Conventional

INTERVENTIONS:
Other: Virtual Reality — Rehabilitation with virtual reality, using Football games, Boxe, Bambolê and Tennis.
  Arms: Virtual Reality Group
Other: Conventional — Stretching exercises in limbs, trunk mobilization in the three planes, balance training in standing position, training of balance reactions and gait training.

SUMMARY:
The aim of this study was to investigate the therapeutic effect of virtual reality associated with conventional physiotherapy on balance during gait and the occurrence of falls in patients after stroke.

DETAILED DESCRIPTION:
Randomized clinical trial conducted with patients of both sexes with hemiparesis after stroke of 18 to 65 years. They excluded those who had less than six months of injury, with sensory or perceptual deficit. Patients included were randomized into two groups, a treatment group, which conducted rehabilitation with virtual reality associated with conventional physical therapy and the control group that performed only conventional physiotherapy. Randomization was done by a computer program in blocks, by a third person, respecting the allocation concealment. After selection and randomization, patients were evaluated at baseline, when they were collected demographic and clinical data, investigated the occurrence of falls in the three months prior to evaluation and rated the balance in motion using the Dynamic Gait Index (DGI). Patients were followed for 20 physiotherapy sessions, visits twice a week for an hour each. The assessment of the balance and the investigation of the occurrence of falls were repeated at the end of treatment, which occurred on average three months after the start of the intervention, by the same examiner, who remained blind to the group that the patient belonged.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes with hemiparesis after stroke of 18 to 65 years.

Exclusion Criteria:

* less than 6 months of injury with sensory or perceptual deficit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index (DGI) | avarage 8 weeks
  Balance during gait in patients after stroke undergoing rehabilitation with virtual reality associated with conventional physiotherapy.

SECONDARY OUTCOMES:
Number of Falls | avarage 8 weeks
  falls in patients after stroke undergoing rehabilitation with virtual reality associated with conventional physiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Fonseca, Principal Investigator — Pedreira, Érika, M.D.